CLINICAL TRIAL: NCT06267716
Title: Comparison of Pericapsular Nerve Block and Iliopsoas Fascial Plane Block Effects on Postoperative Pain and Motor Weakness in Hip Surgery
Brief Title: Pericapsular Nerve Block and Iliopsoas Fascial Plane Block in Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 274-2023
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Hip Fractures; Peripheral Nerve Block
Keywords: iliopsoas plane block; pericapsular nerve group block; Hip Fractures; postoperative pain; motor weakness
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: prospective randomized standardized triple-blind
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants under general anaesthesia and the orthopaedic surgeon responsible for the study will be blinded to the study groups and the specific block procedures. This surgeon will serve as the sole evaluator of postoperative outcomes. Intraoperative results will be recorded by the anaesthesia technician, who is present in the operating room and unaware of the block procedures. Moreover, the data analysis will be conducted before the data are unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block (Active Comparator): Immediately after the insurance of general anaesthesia and LFCN block application, PENG block was performed by the primary investigator (B.C) following proper skin disinfection with the patient in the supine position. Under the guidance of a low-frequency curvilinear ultrasound probe, the iliopubic eminence and the psoas tendon were identified, and local anaesthetic (20 ml 0,375% bupivacaine) was injected between the periosteum and psoas tendon following negative aspiration.
  Interventions: Procedure: PENG block
- IPP block (Experimental): After ensuring aseptic conditions, the low-frequency curvilinear ultrasound probe was transversely placed caudad to the anterior superior iliac spine, then rotated anticlockwise and slid along the inguinal ligament to detect the head of the femur, as described by Nielsen et al. The primary investigator (B.C.) directed the needle tip into the iliopsoas plane between the iliopsoas muscle and iliofemoral ligament through an in-plane approach, and 10 ml of 0,375% bupivacaine was injected.
  Interventions: Procedure: IPB

INTERVENTIONS:
Procedure: PENG block — preoperative ultrasound-guided pericapsular nerve group block
  Arms: PENG block
Procedure: IPB — preoperative ultrasound-guided iliopsoas plane block
  Arms: IPP block

SUMMARY:
This prospective randomized interventional study aims to compare the effects of two peripheral nerve blocks, the periencapsular nerve block (PENG) and iliopsoas block (IPB), on analgesia and motor function after hip surgery.

The main questions it aims to answer are the effectivity of postoperative pain management the preservation of motor movement.

Participants will receive standardized general anesthesia and postoperative PENG or IPB in either Group.

Researchers will compare the total amount of rescue analgesia and numeric rating scale with accompanying evaluating motor function at the same time intervals within 24 hour.

DETAILED DESCRIPTION:
Providing postoperative analgesia after hip joint surgery is essential in ensuring patient recovery and rehabilitation. The blocks that can be used as alternatives in these surgeries have diversified in recent years, and their superiority over each other is being investigated. The aim is to reach a method that provides more effective analgesia, is more practical and does not cause muscle weakness. For this reason, PENG, which has no previous comparative randomized studies, and iliopsoas blocks, which have more recent clinical studies, need to be examined.

All patients received standard general anaesthesia under standard monitoring along with the bispectral index (Medtronic) and nociception level index (NOL, MedaSense). Intubation was performed by administering intravenous (IV) 0,03 mg/kg midazolam 2 mg/kg, propofol (Lipuro, Braun), 2 mcg/kg fentanyl (Talinat, VEM), 0,6 mg /kg rocuronium (Esmeron, Alessandroorsini) followed by 1 MAC sevoflurane (Sevorane, Abbott) in an air-oxygen mixture for maintenance of anaesthesia. All participants received 20 mg tenoxicam and 1 gr paracetamol along with 8 mg dexamethasone before surgical incision as part of multimodal analgesia. All blocks were performed before surgical incision following the induction of general anaesthesia by a single experienced regional anaesthesiologist (B.C.) under ultrasound guidance (Esaote MyLab ™ Seven). Both groups received lateral femoral cutaneous nerve (LFCN) block by using a high-frequency probe to visualize LFCN between sartorius and tensor of fascia lata in line with the inguinal ligament, and 5 ml 0,375 bupivacaine was injected. After applying PENG or IP block in accordance with randomization, the surgery was set to begin after at least 15 minutes of block procedures. The intraoperative analgesic need was supplied by remifentanil infusion (2 mcg/mL) and determined by NOL index level, and a value over 25 for more than one minute was accepted as pain to be treated by increased remifentanil infusion doses. All patients received 8 mg of ondansetron and suggamadex (2 mg/kg) for decurarization before arousal under BIS guidance. From the beginning of acclaimed arousal till the 24th hour, rescue analgesia as tramadol 100 mg (maximum daily dose 400 mg) is applied if NOL is over 25 at the recovery room or NRS over 4 or with the patient's request. The routine analgesia regimen was 1 gram iv paracetamol 6th hourly postoperatively at the orthopaedic ward.

PENG block procedure Immediately after the insurance of general anaesthesia and LFCN block application, PENG block was performed by the primary investigator (B.C) following proper skin disinfection with the patient in the supine position. Under the guidance of a low-frequency curvilinear ultrasound probe, the iliopubic eminence and the psoas tendon were identified, and local anaesthetic (20 ml 0,375% bupivacaine) was injected between the periosteum and psoas tendon following negative aspiration.

IPB procedure After ensuring aseptic conditions, the low-frequency curvilinear ultrasound probe was transversely placed caudad to the anterior superior iliac spine, then rotated anticlockwise and slid along the inguinal ligament to detect the head of the femur, as described by Nielsen et al. The primary investigator (B.C.) directed the needle tip into the iliopsoas plane between the iliopsoas muscle and iliofemoral ligament through an in-plane approach, and 10 ml of 0,375% bupivacaine was injected.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion in this study were those aged 18 to 90 years who had undergone total hip arthroplasty surgery and had an American Society of Anesthesiologists (ASA) Physical Status classification of I to III and body mass index (BMI) between 18 and 30 kg/m2.

Exclusion Criteria:

* Patients were excluded if they had one of the following criteria: refusal to participate, a history of neurological deficits or neuropathy affecting the lower extremity, infection at the site of block application, coagulopathy; allergy to local anaesthetics, epilepsy or treatment with antipsychotics; abuse of alcohol or drugs; previous surgery distorting the anatomy of the inguinal or supra inguinal areas; severe organ dysfunction ( kidney, liver and other); uncooperative patients who fail to respond reliably to verbal pain assessment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
pain scores | postoperative 24 hour
  numeric rating scales as (NRS) which ranges from 0 to 10, where zero represents the absence of pain, and 10 signifies the worst imaginable pain. NRS scores were evaluated at several time points. Prior to data analysis, the primary outcome was revised due to the unexpectedly low incidence of clinically detectable postoperative motor dysfunction observed during trial conduct, which limited its discriminative value. Pain-related outcomes were therefore designated as primary to better reflect clinically meaningful differences between interventions.

SECONDARY OUTCOMES:
postoperative motor block | postoperative 24 hour
  postoperative motor block was assessed using knee extension and hip adduction observed by the blinded orthopedic surgeon. Prior to data analysis, the primary outcome was revised due to the unexpectedly low incidence of clinically detectable postoperative motor dysfunction observed during trial conduct, which limited its discriminative value.
total analgesia, intraoperative | intraoperatively
  intraoperative remifentanil needed guided by nociception level index monitorization. Total intraoperative remifentanil consumption was planned to be recorded under nociception level index guidance. However, due to technical and recording limitations, reliable quantitative remifentanil dose data could not be consistently captured for all participants; therefore, this outcome will not be included in the final comparative analysis.
total rescue analgesia | postoperative 24 hour
  rescue analgesia will be given as tramadol 100 mg if pain scores over 4 or existance of patient request

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, MD, Principal Investigator — Haseki Training and Research Hospital Anesthesiology and Reanimation Department
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jessen C, Brix LD, Nielsen TD, Espelund US, Lund B, Bendtsen TF. Efficacy of iliopsoas plane block for patients undergoing hip arthroscopy: a prospective, triple-blind, randomized, placebo-controlled trial. Reg Anesth Pain Med. 2025 Jan 7;50(1):5-10. doi: 10.1136/rapm-2023-104989. PMID 38050149
- [Background] Yeoh SR, Chou Y, Chan SM, Hou JD, Lin JA. Pericapsular Nerve Group Block and Iliopsoas Plane Block: A Scoping Review of Quadriceps Weakness after Two Proclaimed Motor-Sparing Hip Blocks. Healthcare (Basel). 2022 Aug 18;10(8):1565. doi: 10.3390/healthcare10081565. PMID 36011222